CLINICAL TRIAL: NCT03611049
Title: Improving Cognition and Brain Imagery Through Optimal Vitamin D Supplementation in the Elderly
Brief Title: Improving Functionality in Older People
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator (Dr. Peiris) is retiring
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L18-111
Record Dates: First submitted 2018-05-11; First posted 2018-08-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Two parallel interventions in subjects with vitamin D insufficiency. A low dose vitamin D replacement arm and a high dose vitamin D replacement arm
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Vitamin D intervention (Placebo Comparator): intervention includes 800 IU Vitamin D3 replacement
  Interventions: Dietary Supplement: Low dose Vitamin D3
- High dose Vitamin D intervention (Active Comparator): Intervention includes 5000 IU Vitamin D3 replacement
  Interventions: Dietary Supplement: High dose Vitamin D3

INTERVENTIONS:
Dietary Supplement: High dose Vitamin D3 — High dose arm- 5000IU given daily
  Arms: High dose Vitamin D intervention
Dietary Supplement: Low dose Vitamin D3 — Low dose arm-800 IU given daily
  Arms: Low dose Vitamin D intervention

SUMMARY:
The study will examine if overall functionality of older adults with Vitamin D insufficiency can be improved by optimal Vitamin D replacement over a period of approximately one year. A variety of outcome metrics will be examined including mental and physical parameters

DETAILED DESCRIPTION:
The decline in brain function with aging is costly. The maintenance of optimal brain health is a priority among the elderly. Complex modifiable factors impact brain function such as education level, ongoing use of cognitive skills such as mentoring and social interaction. In most instances, substantial time and effort will be required to improve brain function in the elderly. There is an urgent need for an option that will yield rapid results. Investigator(s) believe intensive Vitamin D replacement presents such a solution.

Emerging scientific information supports an important role for Vitamin D in brain health. Much of this data is based on the association that higher Vitamin D values are linked to better brain function. However, an association does not prove a cause and effect. To prove that Vitamin D values play a causal role in cognition carefully controlled studies are needed. Currently, there are very few controlled interventional studies in the elderly demonstrating that Vitamin D levels can improve brain function. The 25(OH) Vitamin D is the best indicator of Vitamin D status. The normal range for 25(OH) Vitamin D is usually between 30 and 100 ng/ml. Preliminary data indicates that 25(OH) Vitamin D values of greater than 40 ng/ml are needed to improve brain function. Prior Vitamin D studies have used varying replacement protocols and types of Vitamin D such that stable 25(OH) Vitamin D values in the high normal range have rarely been achieved.

Brain Impairment usually occurs gradually in dementia, giving the patient and the provider an option to slow or halt progression of cognitive deterioration. Disruption in the white matter (reflecting the nerve fibers that conduct electric impulses) of the brain as well as reduction in brain volumes are linked to dementia and increasing chances of disability. These white matter abnormalities and reduction in brain volumes are commonly present in the elderly and are closely linked to Vitamin D deficiency. Animal studies using Vitamin D support a benefit to cognition. There is a paucity of carefully controlled clinical trials involving humans using appropriate Vitamin D replacement protocols. However, a few preliminary studies do support a benefit to cognition in humans over a study period ranging from 1-15 months. The present proposal addresses this relative deficiency by conducting a double blind controlled study in the Vitamin D insufficient community dwelling elderly.

The hypothesis is that daily 5000 IU Vitamin D3 will regress or at least prevent progression of white matter abnormalities or shrinking of brain volumes. There are specific anatomical defects in the brain linked to Vitamin D deficiency. These deficits include impaired visual memory and executive (higher brain functions). Investigator(s) will assess brain function by tracking changes in a battery of computerized tests that have been proven reliable in assessing brain function. These changes in computerized testing of brain skills will be matched to changes in brain imaging over the course of the 1 year study. Brain imaging will be done using a 3-Tesla Magnetic Resonance Imaging scan (MRI).

Once the institutional review board approves this study, free living participants (> 65 yrs.) without prior brain disease or dysfunction will be recruited. The participants with Vitamin D insufficiency (25(OH) Vitamin D < 30 ng/ml) will be randomized into two groups. Both participant groups will be treated for 1 year with daily Vitamin D3 supplements. The standard of care group will get 800 IU daily whereas the active group will get 5000 IU daily. Cognitive tests, chemistry profile will be done at baseline and every 4 months for 1 year. The basic chemistry profile (blood work) includes kidney function and calcium levels which also provide safety monitoring. Based on published information, Vitamin D3 doses planned in this study are far below the doses required for toxicity. The brain MRI will be done at baseline, 4 and 12 months.

Additional strengths of this study include a multidisciplinary team with published expertise and experience in Vitamin D replacement, brain and memory function.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling subject (adults) aged between 65 and 89 years of age
* Subject should be ambulatory and living at home
* Subject should be capable of self-care
* Subject should be able to drive an automobile independently and without assistance
* Subject should agree to home visitation by CRI coordinators to assess pill counts or willing to come to TTUHSC for such a visit
* 25(OH) Vitamin D value < 30 ng/ml

Exclusion Criteria:

* Participant unable or unwilling to have follow up for the duration of the study
* Subject that cannot take a daily supplement
* Subject unable to have MRI imaging
* Subject on peritoneal or hemodialysis
* Subject unwilling to have multiple blood draws
* Subject with Sarcoidosis or diseases associated with hypercalcemia
* Subject currently taking supplements containing Vitamin D
* Subject with prior cerebrovascular disease or memory problems
* Subject with prior myocardial infarction or atrial fibrillation or on anticoagulants
* Subject on medications for memory or cognitive issues or mental ill-health
* Subject with life expectancy less than 2 years
* Subject receiving assistance for self-care
* Subject cannot pass motor screening test for valid assessment of cognition
* Subject on medications for Diabetes
* Subject on medication for hypertension

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 1 year
  Muscle strength will be determined by hand grip
Gait speed | 1 year
  Gait speed will be determined by timed walking
Hippocampal and brain volumes | 1 year
  Using a 3 Tesla MRI scanner using FreeSurfer software. Brain volumes are estimated in cubic centimeters and hippocampal volumes are estimated in cubic millimeters
Body composition and regional fat distribution | 1 year
  Body composition will be determined by bioelectrical impedance. Regional fat distribution will be assessed by waist hip ratio. Obesity will be determined through body mass index and percent body fat estimation through bioelectrical impedance
Cognition | 1 year
  Using a battery of tests from Cambridge Cognition. Each test will be given an equal value and a composite cognitive score determined by summation
Quality of Life questionnaire | 1 year
  Quality of life will be determined by SF-36 Questionnaire by Rand

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No